CLINICAL TRIAL: NCT06512415
Title: Comparing 10- Versus 15-mcg Norepinephrine Bolus for Management of Severe Post-spinal Hypotension During Elective Cesarean Delivery: A Randomized, Controlled Trial
Brief Title: 10 Vs.15 mcg Norepinephrine Bolus in Severe Maternal Hypotension During Cesarean Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-421-2022
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Hypotension; Spinal Anesthesia; Cesarean Section
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 mcg group (Active Comparator): patient will receive the study dry once developed severe post-spinal hypotension
  Interventions: Drug: 10 mcg Norepinephrine
- 15 mcg group (Active Comparator): patients will receive the study dry once developed severe post-spinal hypotension
  Interventions: Drug: 15 mcg Norepinephrine

INTERVENTIONS:
Drug: 10 mcg Norepinephrine — The assigned dose (10 mcg) will be diluted with normal saline in a 10-cc syringe
  Arms: 10 mcg group
Drug: 15 mcg Norepinephrine — The assigned dose (15 mcg) will be diluted with normal saline in a 10-cc syringe.
  Arms: 15 mcg group

SUMMARY:
Data regarding the optimum dose of norepinephrine for management of severe maternal hypotension is lacking. A previous report showed that the use of 10-mcg norepinephrine bolus was not superior to the 5-mcg bolus in the management of severe hypotension in addition the incidence of reactive bradycardia and hypertension was comparable in the two doses. Therefore, we hypothesize that using a higher dose of norepinephrine (15 mcg) would increase the success rate of management of severe hypotensive episode.

DETAILED DESCRIPTION:
Upon arrival to the operating room, the patient will be in supine position with left uterine displacement using a wedge below the right buttock. Routine monitoring will be applied (electrocardiography, pulse oximetry, and non-invasive blood pressure monitor). An 18G-cannula will be inserted, and the patients will receive 10 mg metoclopramide. Baseline heart rate and systolic blood pressure will be recorded as the average of three consecutive readings with 2-minutes interval.

Lactated Ringer's solution will be infused at rate of 15 mL/Kg over 10 minutes as a co-load; spinal anesthesia will be achieved by injecting 10 mg of hyperbaric bupivacaine and 20 mcg fentanyl into the subarachnoid space at L3-L4 or L4-L5 interspace using 25G spinal needle.

After subarachnoid block, mothers will be placed in the supine position with left-lateral tilt.

Block success will be assessed after 5 minutes from intrathecal injection of local anesthetic; and will be confirmed if sensory block level is at T4.

The patient would receive the study drug only if she developed severe post-spinal hypotension (defined as systolic blood pressure ≤60% of the baseline reading) as her first hypotensive episode. The management of the hypotensive episode will be considered successful if the systolic blood pressure is > 80% of the baseline within 2 mins of the bolus. If the bolus failed, norepinephrine bolus of 5 mcg will be given.

Any other hypotensive episode (systolic blood pressure <80% of baseline) will be managed with norepinephrine bolus of 5 mcg.

Intraoperative bradycardia (defined as heart rate less than 55 bpm) will be managed by IV atropine bolus (0.5 mg) will be administered.

Fluid administration will be continued up to a maximum of 1.5 liters. An oxytocin bolus (1 IU) will be delivered over five seconds after delivery then infused at a rate of 2.5-7.5 IU/hour.

ELIGIBILITY:
Inclusion Criteria:

* full-term singleton pregnant women
* American society of anesthesiologist II, scheduled for elective cesarean delivery,

Exclusion Criteria:

* Patients with uncontrolled cardiac morbidities (patients with tight valvular lesion, impaired contractility with ejection fraction < 50%, heart block, and arrhythmias),
* hypertensive disorders of pregnancy,
* peripartum bleeding,
* coagulation disorders (patients with INR >1.4 and or platelet count < 80000 /dL) or any contraindication to regional anesthesia,
* baseline systolic blood pressure (SBP) < 100 mmHg

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of successful management of severe post-spinal hypotension | 1 min after spinal anesthesia until 5 min after the delivery
  systolic blood pressure >80% of baseline after drug bolus

SECONDARY OUTCOMES:
time to severe hypotensive episode | 1 min after spinal anesthesia until 5 min after the delivery
  min
reactive bradycardia | 1 min after spinal anesthesia until 5 min after the delivery
  heart rate <55 beat/min
reactive hypertension | 1 min after spinal anesthesia until 5 min after the delivery
  systolic blood pressure >120% of baseline
umbilical blood pH | 5 min after delivery
  umbilical artery sample
Apgar score | 5 min after delivery
  assess Breathing effort, Heart rate, Muscle tone, Reflexes, Skin color, Each category is scored with 0, 1, or 2
systolic blood pressure | baseline, 1 min after spinal anesthesia until 5 min after the delivery
  mmHg
heart rate | baseline, 1 min after spinal anesthesia until 5 min after the delivery
  beat/min

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during the current study are available from the corresponding author upon reasonable request